CLINICAL TRIAL: NCT01646242
Title: Cold Snare Versus Double Biopsy Polypectomy Technique for Removal of Diminutive Colorectal Polyps: a Prospective Randomized Trial
Brief Title: Cold Snare Versus Double Biopsy Polypectomy Technique for Removal of Diminutive Colorectal Polyps
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Chang Kyun Lee, Assistant Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CPP2012
Record Dates: First submitted 2012-07-16; First posted 2012-07-20 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Polyp of Large Intestine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cold snare polypectomy (Experimental)
  Interventions: Procedure: removal of eligible polyps using cold snare polypectomy technique
- Double biopsy polypectomy (Experimental)
  Interventions: Procedure: removal of eligible polyps using double biopsy technique

INTERVENTIONS:
Procedure: removal of eligible polyps using cold snare polypectomy technique — Snare polypectomy using a mini (10 mm open diameter) size electrosurgical snare without application of electrocautery
  Arms: Cold snare polypectomy
Procedure: removal of eligible polyps using double biopsy technique — Cold forceps polypectomy using a standard- capacity forceps with double biopsy technique (two bites per one forceps pass)
  Arms: Double biopsy polypectomy

SUMMARY:
Most of colorectal polyps founded during colonoscopy are diminutive polyps less than 6 mm. However, complete removal of diminutive polyps is required to prevent tumor recurrence and development of potential interval cancers. Currently, a variety of polypectomy techniques such as hot snare, cold snare, and cold forceps polypectomy are frequently used for the removal of diminutive colorectal polyps. In regard to the completeness of polypectomy, there are few data comparing cold snare polypectomy with cold forceps biopsy technique for removal of diminutive (1-5 mm) colorectal polyps. The aim of this study is to compare cold snare polypectomy with cold forceps polypectomy using double biopsy technique for removal of diminutive colorectal polyps.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 20
* Informed consent

Exclusion Criteria:

* Patient undergoing antiplatelets (aspirin, clopidogrel and others) or anticoagulant therapy
* Known existing bleeding tendency (thrombocytopenia or prolonged INR)
* Inflammatory bowel diseases (Crohn's disease, or ulcerative colitis)
* ASA class III or more
* Pregnancy
* Any condition which, in the opinion of the Investigator, places the patient at unacceptable risk if he/she were to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Complete histologic polyp eradication rate | 2 weeks

SECONDARY OUTCOMES:
Time taken for polypectomy (complete visual eradication of each polyp) | 2 weeks
  time from polyp resection to tissue retrieval
Successful tissue retrieval rate of removed tissues | 2 weeks
Rates of adverse events | 4 weeks
  Adverse events include postpolypectomy bleeding and others (polypectomy syndrome or perforation).
Complete visual polyp eradication rate | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chang Kyun Lee, MD, PhD, Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyunghee University Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Church JM. Clinical significance of small colorectal polyps. Dis Colon Rectum. 2004 Apr;47(4):481-5. doi: 10.1007/s10350-003-0078-6. Epub 2004 Mar 4. PMID 14994108
- [Background] Draganov PV, Chang MN, Alkhasawneh A, Dixon LR, Lieb J, Moshiree B, Polyak S, Sultan S, Collins D, Suman A, Valentine JF, Wagh MS, Habashi SL, Forsmark CE. Randomized, controlled trial of standard, large-capacity versus jumbo biopsy forceps for polypectomy of small, sessile, colorectal polyps. Gastrointest Endosc. 2012 Jan;75(1):118-26. doi: 10.1016/j.gie.2011.08.019. PMID 22196811
- [Background] Efthymiou M, Taylor AC, Desmond PV, Allen PB, Chen RY. Biopsy forceps is inadequate for the resection of diminutive polyps. Endoscopy. 2011 Apr;43(4):312-6. doi: 10.1055/s-0030-1256086. Epub 2011 Mar 16. PMID 21412704
- [Derived] Lee CK, Shim JJ, Jang JY. Cold snare polypectomy vs. Cold forceps polypectomy using double-biopsy technique for removal of diminutive colorectal polyps: a prospective randomized study. Am J Gastroenterol. 2013 Oct;108(10):1593-600. doi: 10.1038/ajg.2013.302. Epub 2013 Sep 17. PMID 24042189